CLINICAL TRIAL: NCT03846323
Title: Liberalization of Visiting Policies in ICU for Reducing High Risk of Post-traumatic Stress Disorder (PTSD) in Family Members.
Brief Title: Liberalization of Visiting Policies in ICU for Reducing High Risk of Post-traumatic Stress Disorder
Acronym: OPEN-UNIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: AOM08226
Record Dates: First submitted 2018-12-06; First posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2018-05

CONDITIONS: PTSD in Family Members of ICU Patients
Keywords: Posttraumatic stress disorder (PTSD); ICU; visiting hours policies
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visiting policies: open 24h/24 (Experimental): Visiting policies: 24 hours a day, 7 days a week
  Interventions: Other: Visiting policies: 24 hours a day, 7 days a week
- Restriction of visiting policies (Other): Restriction of visiting policies < 6 hours
  Interventions: Other: Restriction of visiting policies < 6 hours

INTERVENTIONS:
Other: Visiting policies: 24 hours a day, 7 days a week
  Arms: Visiting policies: open 24h/24
Other: Restriction of visiting policies < 6 hours
  Arms: Restriction of visiting policies

SUMMARY:
This was a cluster randomized study of an ICU level intervention to reduce high risk of post-traumatic stress disorder (PTSD) in family members of ICU patients.

Participating ICUs had restrictive visiting policies (i.e., <6 hours/day) before randomization.

After an observational period and a washout period, participating ICUs were randomized either to maintain their visiting policies or to liberalize their visiting policies (24 hours a day, 7 days a week.)

DETAILED DESCRIPTION:
Family members of ICU patients are particularly exposed to anxiety, depressive, acute stress disorder, and posttraumatic stress disorder symptoms (PTSD).

It is currently unknown what type of interventions/ strategies to cope with postintensive care syndrome family would produce the best improvement. Experts suggest that symptoms in family members are potentially amenable to intervention by ICU staff. One intervention to reduce PTSD could be a liberalization of the visiting hours. However, restrictions on visiting hours in the intensive care unit (ICU) are usually adopted worldwide.

ELIGIBILITY:
Inclusion criteria :

Patient and family member > 18 years or older,

* mechanical ventilation expected for more than 48 h and inclusion between day 3 and 5 from the beginning of mechanical ventilation,
* patient having a family member speaking and understanding French, and with the ability to visit his/her relative during the ICU stay,
* patient and his/her relative consenting to participate in the study, or obtention of family consent in case of patient incompetency

Exclusion criteria :

- Patient without family available or family not speaking or understanding French"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1289 (Actual)
Dates: Start 2009-04-18 (Actual); Primary Completion 2013-12-17 (Actual); Study Completion 2018-02-12 (Actual)

PRIMARY OUTCOMES:
Symptoms related to posttraumatic stress disorder (PTSD) | at day-90 from patient's ICU discharge
  Impact event scale (IES). The Impact of Event scale (IES), which assesses symptoms related to post-traumatic stress disorder (PTSD); scores range from 0 (no PTSD-related symptoms) to 75 (severe PTSD-related symptoms).

SECONDARY OUTCOMES:
Beliefs and attitudes of healthcare workers toward visiting hours | 120 days
  Beliefs and Attitudes toward Visitation in ICU Questionnaire (BAVIQ). Beliefs and attitudes of ICU staff members were recorded at the beginning of period 1 (observation period) and at the end of period 2 (intervention period) using a questionnaire named the Beliefs and Attitudes toward Visitation in ICU Questionnaire (BAVIQ). The "Beliefs" questionnaire contains both positively and negatively formulated questions. To calculate an overall score for nurses 'beliefs, we recoded the responses on the negatively formulated questions. Subsequently, we computed the average score over all the belief items. A score of zero corresponded with beliefs that are strongly opposed to open visitation and a score of 4 corresponded with beliefs that are strongly in favor of open visitation.
Family member's needs | At inclusion
  Critical Care Family Needs Inventory (CCFNI) Family needs and satisfaction was measured by a modified version of the Critical Care Family Needs Inventory (CCFNI). The satisfaction score was calculated as the sum of the scores on all items; the smallest possible score was 0 (extreme dissatisfaction) and the highest possible score was 14 (extreme satisfaction).
Family members' symptoms of anxiety and depression | At inclusion and Day-90 from patient's ICU discharge
  Hospital and Anxiety Depression Scale (HADS) The Hospital and Anxiety and Depression Scale (HADS), subscale scores range from 0 (no distress) to 21 (severe distress), HADS subscales scores 5Anxiety and Depression) above 8 were considered to indicate clinically significant symptoms of anxiety or depression.
the proportion of family members with High risk of PTSD occurrence | At day-90 from patients'ICU discharge
  Score IES > 30 points
Patients' symptoms of anxiety and depression | At day-90 from patients'ICU discharge
  Hospital and Anxiety Depression Scale (HADS) The Hospital and Anxiety and Depression Scale (HADS), subscale scores range from 0 (no distress) to 21 (severe distress), HADS subscales scores (Anxiety and Depression) above 8 were considered to indicate clinically significant symptoms of anxiety or depression.
the proportion of patients with High risk of PTSD occurrence | At day-90 from patients'ICU discharge
  Score IES > 30 points

CONTACTS AND LOCATIONS:
Overall Officials: LILA BOUADMA, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: No